CLINICAL TRIAL: NCT06838845
Title: Prospective Observational Study Of Upadacitinib in Ulcerative Colitis in China
Brief Title: An Observational Study to Evaluate Effectiveness and Safety of Upadacitinib in Chinese Adult Participants With Moderate to Severely Active Ulcerative Colitis (UC)
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-085
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label

SUMMARY:
Ulcerative colitis (UC) is a chronic, relapsing, and incurable inflammatory disease of the large intestine. The hallmark clinical symptoms include bloody diarrhea associated with rectal urgency and tenesmus.. This study will assess how effective upadacitinib is in treating UC within a Chinese population.

Upadacitinib is an approved drug for treating UC. Approximately 80 adult participants, who have been prescribed upadacitinib for UC by their physician in accordance with local label, will be enrolled in China.

Upadacitinib will be administered in accordance with the terms of the local marketing authorization, and treatment of participants will be determined solely by the investigator. Participants in the study will be followed for up to 1 year.

There will be no additional burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and only data which are routinely collected during a regular visit will be utilized for this study.

ELIGIBILITY:
Inclusion Criteria:

* Chinese participants meet the diagnosis of moderately to severely active Ulcerative colitis (UC)
* Participants prescribed upadacitinib at discretion of their treating physicians based on sufficient consideration of benefits/risks for patients per local label
* Participant must be an adult (≥ 18 years)
* Participant must provide written authorization to use personal and/or health data prior to the entry into the study

Exclusion Criteria:

* Participant participating in any interventional trials
* Participant with any contraindication to upadacitinib as listed on the local China label
* Participant unwilling or unable to comply with the study requirements, including completion of patient reported outcome questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese adult participants with diagnosis of moderate to severe UC with Tumor Necrosis Factor Inhibitor-Inadequate Responder (TNF-IR) or have contraindications to Tumor Necrosis Factor (TNF) blockers, and commenced on upadacitinib treatment prescribed as part of their routine clinical care at their clinician's discretion according to locally approved label and local treatment prescription recommendations/guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Achievement of clinical response per partial adapted Mayo score. | At Week 8
  Defined as a decrease in Partial Adapted Mayo score of ≥ 1 point and a decrease of ≥ 30% from Baseline, PLUS either a decrease in rectal bleeding sub-score (RBS) of ≥ 1 point or an absolute RBS of ≤ 1.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- China (3):
  - The First Affiliated Hospital, Sun-Yat Sen University /ID# 272997, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 274753, Guangzhou, Guangdong
  - The Second Affiliated Hospital Of Zhengzhou University /ID# 274754, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-085